CLINICAL TRIAL: NCT07288775
Title: Controlled Clinical Trial Between Sleep-Wake Quality and Adjustment of Nocturnal Medical Orders in Hospitalized Patients at Hospital Clinica Nova
Brief Title: Relationship Between Sleep-Wake Quality and Nocturnal Medical Orders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinica Nova (Other)
Responsible Party: Principal Investigator, Maria Elena Romero Ibarguengoitia, Principal Investigator, Hospital Clinica Nova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sleep
Record Dates: First submitted 2025-11-18; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sleep Quality
Keywords: sleep hygine; REM sleep; Non-REM sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Sleep enhancement intervention
- Control (Placebo Comparator)
  Interventions: Behavioral: Standard

INTERVENTIONS:
Behavioral: Sleep enhancement intervention — Adjusted nocturnal medical orders
  Arms: Intervention
Behavioral: Standard — Standard hospital care
  Arms: Control

SUMMARY:
The goal of this randomized controlled clinical trial is to evaluate if the implementation of an adjusted nighttime medical order protocol can improve sleep quality and stabilize physiologic parameters in hospitalized adult patients admitted to general wards.

The main questions it aims to answer are:

Does reducing non-urgent nocturnal medical interruptions increase total sleep time and REM duration? Does improving sleep continuity enhance subjective sleep quality and physiologic stability (heart rate, blood pressure)? Researchers will compare the intervention group (patients under an adjusted nighttime order protocol) with the control group (standard hospital care) to determine whether reorganizing nighttime medical routines improves objective and perceived sleep outcomes.

Participants will:

Wear a Fitbit Sense® device to continuously monitor objective sleep parameters across three hospital nights.

Complete the Pittsburgh Sleep Quality Index (PSQI) at admission and discharge to assess subjective sleep quality.

Undergo standard nighttime vital sign evaluations according to their assigned study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients admitted within the past 24 hours
* Aged 18-65 years
* Hospitalized in the general ward of Hospital Clínica Nova
* Minimum in-hospital stay ≥ 3 days
* Visual Analog Scale for pain < 3
* Glasgow Coma Scale > 13

Exclusion Criteria:

* Visual, hearing, intellectual, or cognitive disability
* History of sleep disorders or obstructive sleep apnea
* Use of antidepressants, anxiolytics, hypnotics, or CNS stimulants
* Hemodynamic instability upon admission or during hospitalization
* Patients transferred from the ICU

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Objetive changes in REM sleep | 3 days
  Change in REM sleep duration (minutes), objectively measured using the Fitbit Sense, after two consecutive nights with reduced nocturnal interruptions compared with one baseline night without modification of medical instructions, and between groups with and without the intervention.
Subjective sleep quality changes | 3 nights
  Sleep-wake quality will be assessed through the Pittsburgh Sleep Quality Index (PSQI), a validated instrument that evaluates subjective sleep quality across seven components. PSQI global scores will be compared between the intervention and control groups to determine whether reducing nocturnal interruptions is associated with improved subjective sleep-wake quality.

SECONDARY OUTCOMES:
Differences in sleep-wake quality between male and female participants | 3 nights
  Sleep-wake quality will be assessed through the Pittsburgh Sleep Quality Index (PSQI), a validated questionnaire that evaluates subjective sleep quality across seven components (sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, daytime dysfunction, and overall sleep quality). PSQI global scores will be compared between male and female participants to determine gender-related differences in sleep-wake quality
Association between sleep-wake quality and participant age | 3 nights
  Sleep-wake quality will be evaluated using the Pittsburgh Sleep Quality Index (PSQI). The association between PSQI global scores and participant age will be analyzed to determine whether increasing age correlates with changes in subjective sleep-wake quality.
Association between sleep-wake quality and body mass index (BMI). | 3 nights
  Sleep-wake quality will be assessed through the Pittsburgh Sleep Quality Index (PSQI). The association between PSQI global scores and body mass index (BMI) will be explored to evaluate whether differences in BMI are related to variations in subjective sleep-wake quality.
Changes in vital signs (heart rate, respiratory rate, body temperature, and oxygen saturation) between the intervention and control groups | 3 nights
  Vital signs-including heart rate, respiratory rate, body temperature, and oxygen saturation-will be monitored using standard clinical measurement devices and/or Fitbit Sense sensor data (as applicable). Changes in these parameters will be compared between the intervention group and the control group to determine whether reducing nocturnal interruptions results in measurable physiologic differences.
Objective changes in NREM sleep | 3 nights
  Change in NREM sleep duration (minutes), objectively measured using the Fitbit Sense, after two consecutive nights with reduced nocturnal interruptions compared with one baseline night without modification of medical instructions. And compared between groups with and without the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinica Nova de Monterrey, San Nicolás de los Garza, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided